CLINICAL TRIAL: NCT06638411
Title: Nocebo Education to Reduce the Potential Unintended Harms of Mental Health Awareness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daria Sandra, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 45738
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: ADHD
Keywords: ADHD; Nocebo Effect; Mental Health Awareness
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be blinded to the study hypotheses and treatment arms, and to the type of intervention they are receiving. Outcome assessors will be blinded to participants' treatment arm assignment and the type of intervention they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADHD information workshop (Experimental)
  Interventions: Behavioral: ADHD information workshop
- ADHD information workshop with nocebo education (Experimental)
  Interventions: Behavioral: ADHD information workshop with nocebo education
- Sleep and dreams workshop (Active Comparator)
  Interventions: Behavioral: Sleep workshop

INTERVENTIONS:
Behavioral: ADHD information workshop — ADHD information workshop that will be delivered by a clinical psychology student in one 30-minute session to a group of participants. The workshop will present information about lesser-known or commonly misdiagnosed ADHD symptoms. To control for the duration of the nocebo module (see the condition below), participants will also learn about sleep and its relevance for maintenance of good cognitive health. At the end, the workshop will involve a writing reflection activity about personal experiences with ADHD symptoms.
  Arms: ADHD information workshop
Behavioral: ADHD information workshop with nocebo education — ADHD information workshop that will be delivered by a clinical psychology student in one 30-minute session to a group of participants. The workshop will present information about lesser-known or commonly misdiagnosed ADHD symptoms, together with a module on nocebo effects and their potential role in worsening symptoms. The nocebo module will describe the current understanding of the role of expectations in creating side effects and elaborate on how this applies to the field of mental health through a series of examples. It will also involve a writing reflection activity about personal experiences with ADHD symptoms, potential for nocebo effect when talking about ADHD symptoms, and ability to apply this information to personal experiences.
  Arms: ADHD information workshop with nocebo education
Behavioral: Sleep workshop — An information workshop about sleep and dream experiences that will be delivered by a clinical psychologist in one 30-minute session to a group of participants. It will be matched on duration, type of content, and engagingness with the experimental sessions.
  Arms: Sleep and dreams workshop

SUMMARY:
This project has two aims. First, the research team will confirm whether providing a mental health awareness workshop poses unintended harms by raising the rate of self-diagnosis (as opposed to a neutral workshop) and causing worsening symptoms in previously healthy young adults over a period of one week. The study will focus on determining this in the context of ADHD, as it includes broad symptoms that overlap with normal experience, is commonly overdiagnosed, and is included in many awareness campaigns for neurodiversity and mental health.

Second, the study will test whether nocebo effect education, or in other words, learning about the nocebo effects, during mental health awareness sessions "inoculates" against them. Simply learning about the role negative expectations play in creating side effects has been shown to reduce nocebo side effects of medications; perhaps, the same applies to mental health.

Researchers will compare the outcome of the ADHD workshop with that of the same workshop but with nocebo information included; both experimental conditions will also be compared to an active control condition. Participants are hypothesised to report the following pattern of symptoms:

ADHD information > ADHD + nocebo education > Control

During the study participants will:

1. Randomize the participants to one of the three workshop conditions to watch
2. Report self-diagnosis score immediately after the workshop and 1 week later.
3. Report symptoms 1 week later.

DETAILED DESCRIPTION:
Rates of mental health problems have risen dramatically in North America and around the world. The high rates of mental health problems led to more mental health awareness efforts on university campuses, in the workplaces, and online. These efforts have greatly destigmatised mental health and increased help seeking across all ages, but may also induce the nocebo effect: it may create negative expectations about one's mental health status and thus paradoxically worsen the very symptoms they try to prevent. Nocebo effect is well known to cause various negative outcomes in medicine, such as worse medication side effects. For instance, when the person takes the drug, she can have negative expectations about having side effects and experience them due to misinterpreting normal but ambiguous physical sensations as the relevant side effects. Mental health awareness campaigns may follow the same pattern: they may reframe normal difficulties that are typical of emerging adulthood as early symptoms of psychiatric disorders, thus exacerbating mental health concerns. Experts are now calling for more balanced approaches to mental health awareness that provide necessary information without causing unintended harms.

This will be a randomized controlled trial designed to evaluate whether mental health awareness induces worsening of symptoms (unintended harms) and whether nocebo education can reduce or inoculate against these. Participants in this study will be recruited from the University of Toronto community and complete the study in small to medium sized groups.

Groups of participants will be assigned to one of the three conditions using block randomisation (in a 1:1:1 ratio). The three conditions will include two experimental conditions and an active control: ADHD information workshop, ADHD information with nocebo education workshop, or a control sleep education workshop. Participants will report their ADHD symptoms and rates of self-diagnosis prior to participating in the workshop, immediately after (self-diagnosis), and at one-week follow-up (both).

ELIGIBILITY:
Inclusion Criteria:

1. No existing diagnosis of ADHD, or history/current diagnosis of any other neurological/psychiatric disorder.
2. Score below 18 on the Adult ADHD Self-Reported Symptom (ASRS) Checklist Screener.
3. No current intake of medication to treat a psychiatric disorder (e.g., antidepressants)
4. Fluent in English;
5. Access to a computer, tablet, or smartphone with internet capability;
6. Normal or corrected-to-normal vision and hearing.

Exclusion Criteria:

1. Diagnosis of ADHD or any other neurological/psychiatric disorder.
2. Active intake of medication.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2024-12-08 (Actual)

PRIMARY OUTCOMES:
Self-reported ADHD symptoms | Change 1 week
  As measured by Adult ADHD Self-Reported Symptom Scale (ASRS), a self-reported scale of ADHD symptoms with a score range of 0-72, with a higher score indicating worse symptoms.
Self-diagnosis with ADHD | Change: Immediate, 1 week
  As measured by one item with a score range from 1 to 5, with a higher score indicating stronger self-diagnosing belief.

SECONDARY OUTCOMES:
Memory Failures | Change, 1 week
  Measured by Memory Failures Scale (MFS), a self-reported scale. The scale ranges in scores from 12-60, where a higher score indicates more failures.
Depressive and Anxiety Symptoms | Change, 1 week
  As measured by the Kessler General Distress Scale (K10). The scale score ranges from 10 to 50, where higher scores indicate more symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Researchers will share anonymised data by depositing it in a data repository (e.g., Open Science Framework).
  We will also provide the statistical analysis plan for the data analysis.
Supporting Information: SAP

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT06638411/Prot_SAP_000.pdf